CLINICAL TRIAL: NCT03230136
Title: Protection During Cardiac Surgery.
Acronym: ProCCard
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 69HCL17_0174
Record Dates: First submitted 2017-07-24; First posted 2017-07-26 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Thoracic Surgery; Cardiopulmonary Bypass
Keywords: Myocardial injury; Ischemia reperfusion; cardiac surgery; cardioprotection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multimodal cardioprotection therapeutic strategy (Experimental)
  Interventions: Other: multimodal cardioprotection strategy
- Traditional anesthetic and therapeutic (Active Comparator): standard anesthetic procedure No intervention (Control).
  Interventions: Other: standard anesthetic procedure

INTERVENTIONS:
Other: multimodal cardioprotection strategy — Multimodal cardioprotection therapeutic strategy will include (1) remote ischemic preconditioning, (2) volatile anesthetic sevoflurane-induced preconditioning, (3) blood glucose control every 30 minutes during cardiac surgery, (4) temporary respiratory acidosis prior to the aortic cross-unclamping and (5) gradual restoration of blood flow after aortic cross-unclamping (gentle reperfusion).
  Arms: Multimodal cardioprotection therapeutic strategy
Other: standard anesthetic procedure — standard anesthetic procedure will include: anesthesia under propofol throughout the cardiac surgery, blood glucose control every 60 minutes, arterial pH maintained at 7.40, theoric blood flow restored at the earliest after aortic cross-unclamping.
  Arms: Traditional anesthetic and therapeutic

SUMMARY:
This trial investigates whether a multimodal cardioprotection per-surgery therapeutic strategy could reduce myocardial injury in patients undergoing cardiac surgery compared to traditional management. The primary endpoint is the AUC (area under the curve) of the hypersensitive troponin I. Blood samples will be collected during the 72 hours following the aortic cross-unclamping. This trial is a French, multicenter, randomized, single-blinded and controlled trial. 210 patients will be enrolled with a clinical follow-up during 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Aortic valve surgery (aortic valve replacement associated or not with coronary artery bypass graft, Bentall surgery or Tirone David surgery)
* Signed informed consent

Exclusion Criteria:

* Emergency surgery
* Redo surgery
* Patient treated with Nicorandil, repaglinid or sulfonylurea 48 hours prior to surgery
* Low cardiac output requiring catecholamine infusion or circulatory assistance prior to surgery
* Severe renal failure: dialysis or glomerular filtration rate < 30 mL/min
* Severe liver failure (spontaneous INR >2)
* Severe respiratory insufficiency (VEMS <40% of predicted value)
* Contra-indication to sevoflurane and propofol
* Myocardial infarction < 7 days
* Severe upper limb arterial disease
* Heparin-induced thrombopenia
* Active infection under antibiotic treatment
* Any other surgery combined with the aortic valve surgery: myotomia of Morrow (hypertrophic myocardiopathy), treatment of heart rhythm disorder, inter-atrial communication closure, mitral valve replacement, tricuspid valve replacement, pulmonary valve replacement.
* Pregnant women
* Currently participating in another trial which may interfere with ProCCard results
* Not benefiting from a social insurance or similar system
* Patient under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-07-03 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of Hypersensitive Troponin I | at 72 hours
  Area under the plasma concentration versus time curve (AUC) of Hypersensitive Troponin I determined for each patient with the serial measurement from of troponin I assays.

SECONDARY OUTCOMES:
Adverse events incidence during the first 30 days following surgery of the multimodal cardioprotection strategy | 30 days
  Adverse events will include death, myocardial infarction, heart failure,arrhythmia requiring medical therapy, neurological disorder such as stroke,respiratory insufficiency, any infectious event, major bleeding requiring transfusion of ≥ 5 U packed red blood cells or surgical intervention or surgical complication
Troponin I serum peak value | 72 hours
  Highest serum value recorded for each patient within 72 hours
Troponin I serum value | 24 hours
  Serum value recorded for each patient within 24 hours
Length of mechanical ventilation | 30 days
Length of stay in intensive care unit (ICU) | 30 days
Length of stay in hospital | 30 days
Index Gravity Score (IGS II, the scoring system measuring the severity of disease for patients admitted to ICU) | 24 hours
  Index Gravity Score provides an estimate of the risk of death: the higher the score is, the higher the risk to die is. The maximum score is 163. The Index Gravity Score includes 17 variables: 12 physiology variables, age, type of admission (scheduled surgical, unscheduled surgical, or medical), and three underlying disease variables (acquired immunodeficiency syndrome, metastatic cancer, and hematologic malignancy).
Number of participants with catecholaminergic support | baseline and 30 days
Dose of catecholaminergic support | baseline and 30 days
3-level version of EQ-5D (EQ-5D-3L) health status score (quality of life score) | Baseline and 30 days
  The 3-level version of EQ-5D consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).It comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'. The VAS can be used as a quantitative measure of health outcome that reflects the patient's own judgement.
number of death | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc FELLAHI, Principal Investigator — Hospices Civils de Lyon
Locations (8):
- France (8):
  - CH Annecy, Annecy
  - Service d'Anesthésie-Réanimation, Hôpital Cardiologique et Pneumologique Louis Pradel, Bron
  - CHU de Caen, Caen
  - service de Chirurgie Cardiaque CHU Gabriel Montpied, Clermont-Ferrand
  - Unité de Réanimation Cardiovasculaire et Thoracique, Hôpital Michallon, Grenoble
  - Clinique de la sauvegarde, Lyon
  - CHU Saint-Etienne, Saint-Etienne
  - Institut Arnault Tzanck - Saint-Laurent du Var, Saint-Laurent-du-Var

REFERENCES:
- [Result] Chiari P, Durand M, Desebbe O, Fischer MO, Lena-Quintard D, Palao JC, Mercier C, Samson G, Varillon Y, Pozzi M, Mewton N, Maucort-Boulch D, Ovize M, Fellahi JL. Multimodal cardioprotective strategy in cardiac surgery (the ProCCard trial): Study protocol for a multicenter randomized controlled trial. Trials. 2019 Sep 11;20(1):560. doi: 10.1186/s13063-019-3638-3. PMID 31511041
- [Result] Chiari P, Mewton N, Maucort-Boulch D, Desebbe O, Durand M, Fischer MO, Lena-Quintard D, Palao JC, Ovize M, Fellahi JL. Multimodal Strategy for Myocardial Protection During Cardiac Surgery: The ProCCard Study. J Am Coll Cardiol. 2021 Feb 16;77(6):827-829. doi: 10.1016/j.jacc.2020.12.020. No abstract available. PMID 33573748